CLINICAL TRIAL: NCT00929838
Title: Telephone Delivered Behavioral Skills Intervention for Blacks With T2DM
Acronym: DM-TBSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leonard Ehianu Egede, Professor & Chair, Department of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: DK81121; R01DK081121 (NIH); R01DK081121-01A1 (NIH); HR18334 (Other: Medical University of South Carolina)
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus, Non-Insulin-Dependent; Diabetes Mellitus, Noninsulin Dependent; Diabetes Mellitus, Type II
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus, Non-Insulin-Dependent; African Americans; Blacks; Randomized Controlled Trial; Controlled Clinical Trial; Behavioral Research; Behavioral Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Information Motivation Behavioral Skills Model

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Diabetes Knowledge/Information Arm (Experimental): Subjects randomized to the diabetes knowledge/information arm will complete 12 diabetes education modules over a 12-week period. The educational materials were developed based on guidelines for diabetes education by the American Diabetes Association. The content is based on the principles of the Adult Learning Theory. The information is designed to be relevant, person centered, and presented in a non-threatening manner. The modules are designed to be delivered via telephone in 10-15 minutes, so that the maximum contact time per telephone call including introduction and closing would not exceed 30 minutes.
  Interventions: Behavioral: Diabetes Knowledge/Information
- Motivation/Behavioral Skills Arm (Experimental): The motivation/behavioral skills intervention consists of patient activation (list of 5 questions to ask their provider at every visit and training on how to ask the questions), patient empowerment (diabetes responsibility contracts, personal goals, and flow charts for patients to record lab results/medications and training on how to use the empowerment tools), and behavioral skills training delivered via telephone lasting 30 minutes every week for 12 weeks. The behavioral skills training will be focused on 4 behaviors - physical activity, diet, medication adherence, and glucose self-monitoring. Guided by subjects' current problem areas and preferences, subjects will be asked to choose 1 of 4 behaviors to focus on every 3 weeks (4 behaviors over 12 weeks).
  Interventions: Behavioral: Motivation/Behavioral Skills
- Combined Intervention Arm (Experimental): The combined intervention group will receive weekly telephone-delivered diabetes knowledge/information, patient activation (list of 5 questions to ask their provider at every visit and training on how to ask the questions), patient empowerment (diabetes responsibility contracts, personal goals, and flow charts for patients to record lab results/medications and training on how to use the empowerment tools), and behavioral skills training delivered via telephone. The behavioral skills training will be focused on 4 behaviors and guided by subjects' current problem areas and preferences, subjects will be asked to choose 1 of 4 behaviors to focus on every 3 weeks. The combined intervention group telephone sessions will last for 30 minutes.
  Interventions: Behavioral: Combined Intervention
- Usual Care Arm (Sham Comparator): The usual care group will receive weekly telephone-delivered general health education lasting 30 minutes for 12 weeks to control for attention. Patients in the usual care group will continue to receive any usual diabetes education provided by the clinic staff; however, they will not receive targeted diabetes knowledge/information, activation, empowerment, or behavioral skills training.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Diabetes Knowledge/Information — This group will receive telephone-delivered diabetes knowledge/information lasting 30 minutes for 12 weeks.
  Arms: Diabetes Knowledge/Information Arm
Behavioral: Motivation/Behavioral Skills — This intervention consists of patient activation, patient empowerment, and behavioral skills training delivered via telephone lasting 30 minutes every week for 12 weeks.
  Arms: Motivation/Behavioral Skills Arm
Behavioral: Combined Intervention — This group will receive all components of the diabetes knowledge/information and the motivation/behavioral skills interventions via telephone lasting 30 minutes every week for 12 weeks.
  Arms: Combined Intervention Arm
Behavioral: Usual Care — This group will receive telephone-delivered general health education lasting 30 minutes for 12 weeks to control for attention and content.
  Arms: Usual Care Arm

SUMMARY:
Blacks or African Americans have greater risk of and are more likely to die from type 2 diabetes (T2DM). Major barriers to effective diabetes care for Blacks include poor diabetes knowledge, self-management skills, empowerment, and perceived control. Few prior studies have tested interventions to address these barriers in combination, especially among Blacks who have the greatest burden of diabetes related complications. This study provides a unique opportunity to address this gap in the literature by testing the efficacy of separate and combined telephone-delivered, diabetes knowledge and motivation/behavioral skills training intervention in high risk Blacks with poorly controlled T2DM. The findings of this study, if successful, will provide new information on how to improve quality of care for diabetes in ethnic minorities and reduce the disproportionate burden of diabetes complications and deaths in this population.

DETAILED DESCRIPTION:
Blacks (African Americans) with Type 2 diabetes (T2DM) have higher prevalence of diabetes, poorer metabolic control, and greater risk for complications and death compared to Whites. Poor outcomes in Blacks with T2DM can be attributed to patient, provider, and health systems level factors. Provider and health system factors account for <10% of variance in major diabetes outcomes. Key differences appear to be at the patient level. Of the patient level factors, consistent differences between Blacks and Whites with T2DM have been found in diabetes knowledge, self-management skills, empowerment, and perceived control. A variety of interventions to improve diabetes self-management have been tested including: 1) knowledge interventions; 2) lifestyle interventions; 3) skills training interventions; and 4) patient activation and empowerment interventions. Most of these interventions have been tested individually, but rarely have they been tested in combination, especially among Blacks who have the greatest burden of diabetes related complications. This study provides a unique opportunity to address this gap in the literature. Using a 2x2 factorial design, this study will test the efficacy of separate and combined telephone-delivered, diabetes knowledge/information and motivation/behavioral skills training intervention in high risk Blacks with poorly controlled T2DM (HbA1c ≥9%). The primary objective is to test the separate and combined efficacy of a telephone-delivered diabetes knowledge/information intervention and motivation/behavioral skills training intervention in improving HbA1c levels in Blacks with T2DM using a 2x2 factorial design. The secondary objectives are: 1) To determine whether patients randomized to the telephone-delivered diabetes knowledge/information intervention, the motivation/behavioral skills training intervention or the combined intervention will have greater improvement in physical activity, diet, medication adherence, and self-monitoring of blood glucose at 12 months of follow-up compared to usual care; and 2) To determine the cost-effectiveness of each telephone intervention separately, and then in combination. The primary outcome is HbA1c level at 12 months of follow-up. The secondary outcomes are cost-effectiveness of each telephone intervention separately, and then in combination, and change in physical activity, diet, medication adherence, and self-monitoring of blood glucose over 12 months of follow-up. The long-term goal of the project is to achieve improvement in diabetes-related outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years
* 2) Clinical diagnosis of T2DM and HbA1c ≥9% at the screening visit
* 3) Self-identified as Black or African American
* 4) Subject must be taking at least one oral medication for diabetes, hypertension, or hyperlipidemia and must be willing to use the MEMS cap and bottle for 12 months
* 5) Subjects must be able to communicate in English
* 6) Subjects must have access to a telephone (landline or cell phone) for the 12 week intervention period

Exclusion Criteria:

* 1) Mental confusion on interview suggesting significant dementia
* 2) Participation in other diabetes clinical trials
* 3) Alcohol or drug abuse/dependency
* 4) Active psychosis or acute mental disorder
* 5) Life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2008-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, MD, MS, Principal Investigator — Medical University of South Carolina (MUSC)
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Egede LE, Strom JL, Durkalski VL, Mauldin PD, Moran WP. Rationale and design: telephone-delivered behavioral skills interventions for Blacks with Type 2 diabetes. Trials. 2010 Mar 29;11:35. doi: 10.1186/1745-6215-11-35. PMID 20350322
- [Result] Egede LE, Williams JS, Voronca DC, Gebregziabher M, Lynch CP. Telephone-Delivered Behavioral Skills Intervention for African American Adults with Type 2 Diabetes: A Randomized Controlled Trial. J Gen Intern Med. 2017 Jul;32(7):775-782. doi: 10.1007/s11606-017-4023-0. Epub 2017 Mar 23. PMID 28337686
- See also: Protocol Paper — http://www.trialsjournal.com/content/11/1/35
- See also: Primary Outcomes Paper — https://pubmed.ncbi.nlm.nih.gov/28337686/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetes Knowledge/Information Arm | Motivation/Behavioral Skills Arm | Combined Intervention Arm | Usual Care Arm
Started | 63 | 65 | 63 | 64
Completed | 53 | 56 | 53 | 55
Not Completed | 10 | 9 | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Knowledge/Information Arm | Motivation/Behavioral Skills Arm | Combined Intervention Arm | Usual Care Arm | Total
Number analyzed (Participants) | 63 | 65 | 63 | 64 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 51 | 48 | 52 | 199
  >=65 years | 15 | 14 | 15 | 12 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 30 | 31 | 114
  Male | 35 | 40 | 33 | 33 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 63 | 65 | 63 | 64 | 255
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) at 12 Months Post Randomization
Time Frame: 12-months post randomization
Population: Final analysis used baseline A1c analysis of covariance for differences in levels of A1c between the treatment groups at 12months with baseline A1c as covariate.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Diabetes Knowledge/Information Arm | Motivation/Behavioral Skills Arm | Combined Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 63 | 65 | 63 | 64
percentage of glycosylated hemoglobin | 9.3 (1.8) | 9.2 (2.1) | 9.2 (1.9) | 9.5 (2.5)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Diabetes Knowledge/Information Arm | Motivation/Behavioral Skills Arm | Combined Intervention Arm | Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/65 | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/65 | 0/63 | 0/64
Other Adverse Events (participants affected / at risk) | 0/63 | 0/65 | 0/63 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2009-02-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT00929838/Prot_000.pdf